CLINICAL TRIAL: NCT01317758
Title: A Randomized, Double-Blinded, Controlled, Phase I Study in Healthy Adults to Assess the Safety, Reactogenicity, and Immunogenicity of Intramuscular Subvirion Inactivated Monovalent Influenza A/H5N1 Virus Vaccine Administered at Different Dose Levels Given With and Without AS03 Adjuvant
Brief Title: H5N1 Mix and Match With AS03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-0017; N01AI80057C
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Influenza
Keywords: influenza, vaccine, H5N1
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — AS03 adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Group 6 (Placebo Comparator): Two doses of sanofi H5N1 antigen 15 mcg plus PBS diluent
  Interventions: Other: Phosphate Buffered Saline (PBS) diluent; Biological: Sanofi H5N1 Antigen
- Group 5 (Placebo Comparator): Two doses of sanofi H5N1 antigen 7.5 mcg plus PBS diluent
  Interventions: Other: Phosphate Buffered Saline (PBS) diluent; Biological: Sanofi H5N1 Antigen
- Group 4 (Placebo Comparator): Two doses of sanofi H5N1 antigen 3.75 mcg plus Phosphate Buffered Saline (PBS) diluent
  Interventions: Other: Phosphate Buffered Saline (PBS) diluent; Biological: Sanofi H5N1 Antigen
- Group 3 (Experimental): Two doses of sanofi H5N1 antigen 15 mcg plus GSK AS03 adjuvant
  Interventions: Drug: AS03 Adjuvant; Biological: Sanofi H5N1 Antigen
- Group 1 (Experimental): Two doses of sanofi H5N1 antigen 3.75 mcg plus GSK AS03 adjuvant
  Interventions: Drug: AS03 Adjuvant; Biological: Sanofi H5N1 Antigen
- Group 2 (Experimental): Two doses of sanofi H5N1 antigen 7.5 mcg plus GSK AS03 adjuvant
  Interventions: Drug: AS03 Adjuvant; Biological: Sanofi H5N1 Antigen

INTERVENTIONS:
Drug: AS03 Adjuvant — Adjuvant/diluent manufactured by GlaxoSmithKline (GSK)
  Arms: Group 1; Group 2; Group 3
Other: Phosphate Buffered Saline (PBS) diluent — Placebo/diluent provided by sanofi pasteur
  Arms: Group 4; Group 5; Group 6
Biological: Sanofi H5N1 Antigen — Subvirion inactivated monovalent influenza A/H5N1 (Hemagglutinin (HA) of A/Indonesia/05/2005) virus vaccine manufactured by sanofi pasteur, at 2 doses levels 21 days apart, administered at 3.75, 7.5, or 15mcg, with either AS03 adjuvant or PBS.

SUMMARY:
Approximately 216, and up to 240, healthy males and non-pregnant females, 18 to 49 years old, inclusive, will be enrolled over a 5-month period into this multicenter, randomized, double-blinded, controlled Phase I study. Subjects who meet the entry criteria for the study and provide informed consent will be randomized 2:1 between adjuvanted and unadjuvanted vaccine and placed into one of 6 groups (see table) to receive two doses of an intramuscular subvirion inactivated monovalent influenza A/H5N1 virus vaccine at 3.75, 7.5, or 15 mcg given with the adjuvant AS03 or diluent (N=216, up to 240). All eligible subjects will receive 2 doses separated by approximately 21 days.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, controlled, Phase I study in healthy male and non-pregnant female subjects, 18 to 49 years old, inclusive, designed to assess the safety, reactogenicity, and immunogenicity of an intramuscular subvirion inactivated monovalent influenza A/H5N1 (HA of A/Indonesia/05/2005) virus vaccine manufactured by sanofi pasteur administered at different dosage levels (3.75, 7.5 or 15 mcg) given with the AS03 adjuvant manufactured by GSK or PBS diluent.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for study entry and Dose 1:

* Are males or non-pregnant females between the ages of 18 and 49 years, inclusive.
* Women of childbearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for >/=1 year) must agree to practice adequate contraception (that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms or diaphragms with spermicide or foam, intrauterine devices, and licensed hormonal methods) during the study for at least 30 days following the last vaccination. Adherence to contraceptive method will be captured on the appropriate case report form (CRF).
* Are in good health, as determined by vital signs (oral temp, pulse and blood pressure), medical history and complete physical examination (without genital and rectal exam) to ensure no existing chronic medical diagnoses or conditions are present.
* ESR less than 30 mm per hour.
* For women of childbearing potential, negative urine or serum pregnancy test within 24 hours prior to the first vaccination.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Inclusion Criteria for Dose 2:

* Have received the first dose of study vaccine.
* For women of childbearing potential, negative urine or serum pregnancy test within 24 hours prior to the second vaccination. Adherence to contraceptive method will be captured on the appropriate case report form (CRF).

Exclusion Criteria:

Exclusion Criteria for study entry and Dose 1:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol-9, thimerosal and chicken protein), or allergy to squalene-based adjuvants.
* Women who are breastfeeding or plan to breastfeed at any given time from the first vaccination until 30 days after the last vaccination.
* Have long term use (defined as taken for 2 weeks or more in total at any time during the past 2 months) of high dose oral or parenteral glucocorticoids (high dose defined as prednisone >/= 20 mg total daily dose, or equivalent dose of other glucocorticoids); or highdose inhaled steroids (high dose defined as >800 mcg/day of beclomethasone dipropionate or equivalent);or systemic corticosteroids of any dose within the past 4 weeks.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
* Hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* Receiving systemic, prescription medications for the treatment of chronic medical conditions, unless such use is on a PRN (as needed) basis only. Non-PRN use of systemic, over-the-counter medications and PRN systemic, prescription medication may be allowed if, in the opinion of the investigator, they pose no additional risk to subject safety or assessment of immunogenicity/reactogenicity. Note: Topical, nasal, and inhaled medications; vitamins; and contraceptives are also permitted.
* Received pre-medication with analgesic or antipyretic agents in the 6 hours prior to first vaccination, or planned medication with analgesic or antipyretic in the week following first vaccination. This criterion should not preclude subjects receiving such medication if the need arises. However, pre-medication is to be discouraged.
* Received immunoglobulin or other blood products (with exception of Rho D immune globulin) within the 3 months prior to the first vaccination.
* Received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to the first vaccination or plan receipt of such vaccines within 42 days following the first vaccination. This is inclusive of licensed seasonal influenza vaccines.
* Have an acute or chronic medical condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would render vaccination unsafe, would interfere with the evaluation of responses or is not generally seen in "normal, healthy subjects".
* Have a history of severe reactions following previous immunization with contemporary influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than or equal to 100.4 degrees F, within 3 days prior to the first vaccination.
* Pulse is less than 40 bpm or greater than 100 bpm. An ECG documenting only sinus bradycardia is required for pulses less than 50 bpm.
* Systolic blood pressure is less than 90 mm Hg or greater than 140 mm Hg.
* Diastolic blood pressure is less than 60 mm Hg or greater than 90 mmHg.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to the first vaccination or expects to receive an experimental agent, other than from participation in this study, during the 13-month study period.
* Are participating or plan to participate in another clinical trial with a licensed product during the 13-month study period.
* Have any condition that would, in the opinion of the site principal investigator or appropriate sub-investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in an influenza A/H5 vaccine study in the past in a group receiving vaccine (does not apply to documented placebo recipients) or have a history of A/H5 infection prior to enrollment.
* Have known active HIV, Hepatitis B, or Hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Plan to travel outside the U.S. in the time between the first vaccination and 42 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the site principal investigator or appropriate sub-investigator believes may interfere with successful completion of the study.

Exclusion Criteria for Dose 2:

* Women who are breastfeeding or plan to breastfeed at any given time from the first vaccination until 30 days after the last vaccination.
* Other than from participation in this study, received an experimental agent (vaccine, drug, biologic, device, blood product, or medication), since receipt of Dose 1, or expects to receive an experimental agent during the 13-month study period.
* Are participating/have participated, since receipt of Dose 1, or plan to participate in another clinical trial with a licensed product during the 13-month study period.
* Use of anticancer chemotherapy or radiation therapy (cytotoxic), new diagnosis of an active malignancy, or is immunosuppressed as a result of an underlying illness or treatment since receipt of Dose 1.
* Use of high dose oral or parenteral glucocorticoids (high dose defined as prednisone >/= 20 mg total daily dose or equivalent dose of other glucocorticoids); or high-dose inhaled steroids (high dose defined as > 800 mcg/day of beclomethasone dipropionate or equivalent); or systemic corticosteroids of any dose for 2 weeks or more in total since receipt of Dose 1. Those patients who have received >/= 6-13 days of steroids, within the past 21 days will require at least 14 days off of steroids prior to administration of the second dose of vaccine - see Section 10.3.3. Under 6 days of steroids, no deferral of the second dose of vaccine is needed.
* Received immunoglobulin or other blood products (with exception of Rho D immune globulin) since receipt of Dose 1.
* Received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to the second vaccination or plan receipt of such vaccines within 21 days following the second vaccination. This is inclusive of licensed seasonal influenza vaccines.
* Have new diagnosis of chronic medical disease or chronic medical condition since receipt of Dose 1 that, in the opinion of the site principal investigator or appropriate sub-investigator, would render vaccination unsafe, would interfere with the evaluation of responses or is not generally seen in "normal, healthy subjects".
* Received systemic, prescription medications for the treatment of chronic medical conditions, unless such use is on a PRN (as needed) basis only since receipt of Dose 1. Non-PRN use of systemic, over-the-counter medications and PRN systemic, prescription medication may be allowed if, in the opinion of the investigator, they pose no additional risk to subject safety or assessment of immunogenicity/reactogenicity. Note: Topical, nasal, and inhaled medications; vitamins; and contraceptives are also permitted.
* Received pre-medication with analgesic or antipyretic agents in the 6 hours prior to second vaccination, or planned medication with analgesic or antipyretic in the week following second vaccination. This criterion should not preclude subjects receiving such medication if the need arises. However, pre-medication is to be discouraged.
* Hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others since receipt of Dose 1.
* New occurrence or new awareness of Guillain-Barré Syndrome since receipt of Dose 1.
* Any unresolved or continuing solicited or unsolicited Grade 2 or greater severity adverse events, including reactogenicity events, that have occurred since receipt of Dose 1 without a clear, alternative etiology. Unresolved or continuing Grade 1 adverse events are permissible unless, in the opinion of the site principal investigator or appropriate sub-investigator, they would render vaccination unsafe, would interfere with the evaluation of responses or are not generally seen in "normal, healthy subjects".
* Grade 2 or greater severity clinical safety lab values (according to the toxicity table, Section 11.1.1.2) that do not return to Grade 1 or less prior to the second vaccination. If the clinical safety lab values return to Grade 1 or less, vaccination should be rescheduled within the acceptable window for the second vaccination - see Section 10.3.3. Subjects who experienced a Grade 3 or above clinical safety laboratory adverse event since receipt of Dose 1 should be excluded from receipt of second vaccination. Subjects who had a Grade 3 or above clinical safety laboratory adverse event prior to first vaccination will be evaluated by the site principal investigator and DMID Medical Monitor to determine receipt of second vaccination.
* Have an acute illness, including an oral temperature greater than or equal to 100.4 degrees F, within 3 days prior to the second vaccination. Vaccination of subjects should be deferred until acute illness, including an oral temperature greater than or equal to 100.4 degrees F, has resolved. If resolution occurs, vaccination should be rescheduled within the acceptable window for the second vaccination - see Section 10.3.3.
* Emergence of Grade 2 or greater severity signs or symptoms since receipt of Dose 1 that could confound or confuse assessment of vaccine reactogenicity.
* Any new clinical findings since receipt of Dose 1, which in the opinion of the site principal investigator or appropriate sub-investigator, would compromise the safety of the subject or would interfere with the evaluation of responses or successful completion of the study.
* Plan to travel outside the U.S. in the time between the second vaccination and 21 days following the second vaccination.
* Subject refuses further vaccination. Subjects who do not receive the second vaccination will be asked to return for safety assessments and for scheduled venous blood sample collections for clinical safety laboratory and immunogenicity evaluations and will be followed for the duration of the study - see the protocol-specific Manual of Procedures (MOP) for further details.
* Subject withdraws consent. The subject may withdraw their consent for study participation at any time and for any reason, without penalty.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: Geometric mean titer (GMT) of HAI antibody, subjects with HAI antibody titer 1:40 or greater, and frequency of 4-fold or greater HAI antibody increase against A/H5N1 vaccine in each group 21 days following 2nd vaccine dose (approx Day 42) | Day 42
Safety/Tolerability: Occurrence of solicited local and systemic reactogenicity in the 8 days (Day 0-7) after each vaccination. | Day 0 through Day 7 after each vaccination
Safety/Tolerability: Occurrence of vaccine-associated serious adverse events (SAEs) and clinical safety laboratory adverse events (AEs) from the time of first vaccination through 13 months after the first vaccination. | From time of 1st vaccination through 13 months

SECONDARY OUTCOMES:
GMT of neutralizing antibody (NA), proportion of subjects with a serum NA titer of 1:40 or greater, and frequency of 4-fold or greater increases of NA against A/H5N1 virus vaccine in each group 21 days following 2nd dose of vaccine (approximately Day 42) | Day 42

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington

REFERENCES:
- [Derived] Chen WH, Jackson LA, Edwards KM, Keitel WA, Hill H, Noah DL, Creech CB, Patel SM, Mangal B, Kotloff KL. Safety, Reactogenicity, and Immunogenicity of Inactivated Monovalent Influenza A(H5N1) Virus Vaccine Administered With or Without AS03 Adjuvant. Open Forum Infect Dis. 2014 Oct 8;1(3):ofu091. doi: 10.1093/ofid/ofu091. eCollection 2014 Dec. PMID 25734159